CLINICAL TRIAL: NCT05378269
Title: Phase 1/2 Study of Intravaginal Tamoxifen (DARE-VVA1): Randomized, Double-blind, Placebo-controlled Study of Safety, Pharmacokinetics and Pharmacodynamics in Postmenopausal Participants With Moderate to Sever Vulvar and Vaginal Atrophy
Brief Title: Study of Intravaginal Tamoxifen in PostMenopausal Women With VVA
Acronym: DARE-VVA1
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Daré Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: DARE-VVA-001
Record Dates: First submitted 2022-05-02; First posted 2022-05-18 (Actual); Results first posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-07

CONDITIONS: Vulvar Atrophy
MeSH Terms: interventions — Tamoxifen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Placebo (Placebo Comparator): Vaginal insert
  Interventions: Other: Placebo
- DARE-VVA1 1mg (Experimental): vaginal insert
  Interventions: Drug: Tamoxifen
- DARE-VVA1 5mg (Experimental): vaginal insert
  Interventions: Drug: Tamoxifen
- DARE-VVA1 10mg (Experimental): vaginal insert
  Interventions: Drug: Tamoxifen
- DARE-VVA1 20mg (Experimental): vaginal insert
  Interventions: Drug: Tamoxifen

INTERVENTIONS:
Drug: Tamoxifen — Tamoxifen vaginal insert
  Arms: DARE-VVA1 10mg; DARE-VVA1 1mg; DARE-VVA1 20mg; DARE-VVA1 5mg
Other: Placebo — Placebo vaginal insert
  Arms: Placebo

SUMMARY:
The purpose of the study is to study the safety, PK and PD of Intravaginal Tamoxifen on postmenopausal women with vulvar vaginal atrophy.

ELIGIBILITY:
Inclusion Criteria:

* 1. Women aged 40-75 (inclusive).

  2. Postmenopausal women with a body mass index between 18 and 34 kg/m2, inclusive.

  3. Postmenopausal, defined as 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum follicle-stimulating hormone levels > 40 mIU/mL or 6 weeks post-surgical bilateral oophorectomy.

  4. Have moderate to severe VVA as determined by self-assessment of the following symptoms (as none, mild, moderate, or severe), with at least 1 symptom reported as moderate or severe: vaginal dryness; vaginal and/or vulvar irritation/itching; dysuria; vaginal pain with sexual activity (dyspareunia); vaginal bleeding associated with sexual activity (presence versus absence).

  5. Women who currently have vaginal intercourse or other sexual activity (masturbation, etc.) at least once a month (with or without a partner), or who had intercourse or other sexual activity at least once a month in the past, but later decreased sexual activity due to excessive pain or vaginal dryness. Participants must be willing to engage in vaginal intercourse or other sexual activity (masturbation, etc.) at least 1 time between Days 49-56 of the clinical study.

  6. Participants, upon pelvic examination with speculum examination, must have a normal-appearing vulva other than atrophic changes, normal-appearing cervix other than atrophic changes (i.e., cervical stenosis and/or flushness with the vaginal wall) and normal-appearing vagina (without erosions, ulcerations, scarring, or evidence of dermatoses) other than atrophic changes (loss of ruggae, mucosal pallor, mucosal dryness, mucosal petechiae).

  7. Have an intact uterus and no prior history of endometrial ablation.

  8. Vaginal cellular cytology with ≤ 5% superficial cells.

  9. Vaginal pH > 5 at Screening Visit.

  10. Endometrial thickness ≤ 4 mm on transvaginal ultrasound.

  11. Current on all recommended screening and management requirements for cervical cancer.

  12. Normal mammogram report within 2 years of screening.

  13. Normal manual breast examination by investigator at baseline.

  14. Baseline hematology, clinical chemistry, urinalysis, prothrombin time/partial thromboplastin time (PT/PTT) and viral serologies for human immunodeficiency virus (HIV), hepatitis C virus (HCV), and hepatitis B surface antigen (HBsAg) all within normal limits OR accepted by the investigator and medical monitor as not clinically significant.

  15. Normal 12-lead electrocardiogram (ECG).

  16. Able to read, understand, and provide written informed consent and applicable data protection authorization after the nature of the study has been fully explained, and must be willing to comply with all study requirements.

  17. Willing and able to correctly and independently complete all study procedures.

Exclusion Criteria:

1. A history of or physical examination finding for any significant cardiovascular, renal, pulmonary, neurological and hepatic diseases preventing compliance with this study.
2. A medical history of or use of anticoagulant drugs to treat or prevent coagulopathies, thrombophilia or thromboembolic disease (deep vein thrombosis, pulmonary or systemic embolism, stroke, or transient ischemic attack).
3. Uncontrolled hypertension (either systolic > 180 mmHg or diastolic > 105 mmHg), treatment with Class 1 antiarrhythmics or digitalis, history of congestive heart failure (New York Heart Association [NYHA] > Class I), or myocardial infarction within 12 months.
4. Abnormal cervical screening test within 2 years of screening. Participant can have atypical squamous cells of undetermined significance if human papilloma virus-negative.
5. History of or current endometrial pathology: hyperplasia, carcinoma and/or polyp (prior history of a benign endometrial polyp with no current evidence of polyp is acceptable).
6. A medical history of breast cancer within 5 years of screening. Participants with a history of breast cancer more than 5 years prior to screening are considered eligible if their disease was node-negative, nonmetastatic, and if all treatment with aromatase inhibitors (AIs) or SERMs was completed at least 6 months prior to screening.
7. A medical history of malignant melanoma.
8. Any cancer (except nonmelanomatous skin cancer) diagnosed less than 5 years prior to the Screening Visit.
9. A medical history of undiagnosed vaginal bleeding.
10. A known or suspected estrogen-dependent neoplasia.
11. Previous radiation treatment to the pelvis.
12. Women who have previously reported an unsatisfactory outcome from a vaginal hormone therapy for VVA.
13. Known hypersensitivity to any ingredients in DARE-VVA1.
14. Use of vaginal hormonal products (rings, creams, gels, tablets, capsules) within 4 weeks prior to Day 1.
15. Use of transdermal estrogen or transdermal estrogen/progestin products within 4 weeks prior to Day 1.
16. Use of oral estrogen and/or progestin therapy within 8 weeks prior to Day 1.
17. Use of intrauterine progestin therapy within 8 weeks prior to Day 1.
18. Use of progestin implants or estrogen-alone injectable drug therapy within 12 weeks prior to Day 1.
19. Administration of estrogen pellet therapy or progestin injectable drug therapy within 6 months prior to Day 1.
20. Use of thyroid hormone replacement therapy unless the participant is on a stable dose for > 6 months, and participant is euthyroid based on a normal, sensitive immunoassay for thyroid-stimulating hormone (TSH).
21. Use of SERMs or AIs within 6 months prior to screening.
22. Use of anabolic or other steroids (including hormonal creams such as testosterone) within 4 weeks prior to Day 1.
23. Use of corticosteroids, > 5 mg/day prednisone or equivalent, for more than 4 weeks within 4 weeks prior to Day 1.
24. Participants with any self-reported active sexually transmitted disease and/or evidence of infection (including bacterial vaginosis) on vaginal examination by the investigator.
25. Participants with a urinary tract infection during screening as assessed by urine dipstick test with abnormal test findings (any positive result for leukocytes AND any positive result for nitrites).
26. Presence of clinically significant uterine fibroids.
27. Evidence of current alcohol or drug abuse in the past 60 days, including a positive result from the urine drugs of abuse or alcohol screen, or history of drug or alcohol dependence in the last 2 years, as assessed by the investigator. Alcohol abuse is defined as greater than 14 standard units/week for females, and drug abuse is defined as known psychiatric or substance abuse disorder that would interfere with participation with the requirements of this study, including current use of any illicit drugs. Use of medical cannabis is not exclusionary.
28. Participation in any other investigational drug or device trial in which administration of an investigational study drug/device occurred within 30 days or placement of a non-drug eluting medical device within 15 days prior to the Screening Visit (Visit 1).
29. In the opinion of the investigator, participant has any disorder or finding that might interfere with the conduct of the study.

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-11-22 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2023-03-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - PARC Clinical Research, Adelaide, Southern Australia
  - Keogh Institute for Medical Research, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: No
A decision has not yet been made on when or what IPD to share when available.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | DARE-VVA1 1mg | DARE-VVA1 5mg | DARE-VVA1 10mg | DARE-VVA1 20mg
Started | 4 | 3 | 4 | 3 | 3
Completed | 3 | 3 | 2 | 3 | 3
Not Completed | 1 | 0 | 2 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | DARE-VVA1 1mg | DARE-VVA1 5mg | DARE-VVA1 10mg | DARE-VVA1 20mg | Total
Number analyzed (Participants) | 4 | 3 | 4 | 3 | 3 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 1 | 4 | 2 | 2 | 12
  >=65 years | 1 | 2 | 0 | 1 | 1 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (5.38) | 65.7 (1.53) | 59.3 (2.99) | 57.7 (8.08) | 61.3 (4.16) | 60.9 (4.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 4 | 3 | 3 | 17
  Male | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 3 | 4 | 3 | 3 | 17
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 4 | 3 | 4 | 3 | 3 | 17
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Australia | 4 | 3 | 4 | 3 | 3 | 17
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 25.03 (5.287) | 26.04 (4.869) | 26.58 (5.486) | 24.67 (2.219) | 23.70 (3.676) | 25.27 (4.151)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Treatment Emergent Adverse Events
Description: to evaluate the safety and tolerability of DARE-VVA1 by intravaginal administration
Time Frame: 56 days
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | DARE-VVA1 1mg | DARE-VVA1 5mg | DARE-VVA1 10mg | DARE-VVA1 20mg
Number analyzed (Participants) | 4 | 3 | 4 | 3 | 3
Participants | 3 | 2 | 4 | 3 | 3

2. Primary Outcome: Concentration of Tamoxifen in Serial Plasma Collections (Cmax)
Description: to determine the plasma concentrations of tamoxifen after intravaginal administration
Time Frame: 56 days
Population: Placebo users were not using Tamoxifen so a correlation between Tamoxifen and vaginal pH was not performed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Placebo | DARE-VVA1 1mg | DARE-VVA1 5mg | DARE-VVA1 10mg | DARE-VVA1 20mg
Number analyzed (Participants) | 4 | 3 | 2 | 3 | 3
ng/mL | 0 (0) | 0.181 (32.21) | 1.93 (46.62) | 3.29 (12.01) | 5.50 (31.54)

3. Secondary Outcome: Evaluation of Vaginal Cytology
Description: to analyze the change from baseline to end of study of percentage of parabasal cells
Time Frame: 56 days
Population: We were looking at a correlation between Tamoxifen and parabasal cells. Placebo users were not exposed to Tamoxifen.
Measure: Mean (Full Range); unit: % parabasal cells
Arm/Group | Placebo | DARE-VVA1 1mg | DARE-VVA1 5mg | DARE-VVA1 10mg | DARE-VVA1 20mg
Number analyzed (Participants) | 4 | 3 | 2 | 3 | 3
% parabasal cells | 0 [0 to 0] | -12.0 [-15 to -5] | -22.5 [-45 to 0] | -69.0 [-98 to -61] | -94.0 [-100 to -04]

4. Secondary Outcome: Evaluation of Vaginal pH
Description: to analyze preliminary efficacy and pharmacodynamics of DARE-VVA1 by looking at change in baseline of vaginal pH from Day 1 to Day 56
Time Frame: 56 days
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Placebo | DARE-VVA1 1mg | DARE-VVA1 5mg | DARE-VVA1 10mg | DARE-VVA1 20mg
Number analyzed (Participants) | 3 | 3 | 2 | 3 | 3
pH | -0.3 (0.95) | -0.3 (0.31) | -0.3 (0.42) | -0.3 (0.70) | -0.7 (0.72)

5. Secondary Outcome: Evaluation of Vaginal Cytology
Description: to analyze the change from baseline to end of study of percentage of superficial cells
Time Frame: 56 days
Population: We were looking at a correlation between Tamoxifen and superficial cells. Placebo users were not exposed to Tamoxifen.
Measure: Mean (Full Range); unit: % superficial cells
Arm/Group | Placebo | DARE-VVA1 1mg | DARE-VVA1 5mg | DARE-VVA1 10mg | DARE-VVA1 20mg
Number analyzed (Participants) | 4 | 3 | 4 | 3 | 3
% superficial cells | 0 [0 to 0] | -3.0 [-4 to -2] | 8.5 [2 to 15] | 6.0 [1 to 14] | 52.3 [18 to 85]

6. Other Pre Specified Outcome: Collection of Menopause-specific Quality of Life (MENQOL) Questionnaire
Description: to analyze the impact of DARE-VVA1 on quality of life following treatment evaluated by total questionnaire score; looking for a decreased in total score.
Time Frame: 56 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 56 days
Arm/Group | Placebo | DARE-VVA1 1mg | DARE-VVA1 5mg | DARE-VVA1 10mg | DARE-VVA1 20mg
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3 | 0/4 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3 | 0/4 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 3/4 | 2/3 | 4/4 | 3/3 | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=4) | DARE-VVA1 1mg (N=3) | DARE-VVA1 5mg (N=4) | DARE-VVA1 10mg (N=3) | DARE-VVA1 20mg (N=3)
Vulvovaginal discomfort (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Vulvovaginal pruritis (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Genital rash (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Postmenopausal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal erythema (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study enrollment proved difficult and lead to small numbers of subjects analyzed per arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI is not able to publish study data without prior approval from Sponsor.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-04): https://cdn.clinicaltrials.gov/large-docs/69/NCT05378269/Prot_SAP_000.pdf